CLINICAL TRIAL: NCT02099123
Title: A Study of STAtins for Reducing Events in the Elderly (STAREE)
Brief Title: A Clinical Trial of STAtin Therapy for Reducing Events in the Elderly (STAREE)
Acronym: STAREE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); National Heart Foundation, Australia (Other)
Responsible Party: Principal Investigator, Sophia Zoungas, Professor Sophia Zoungas, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NHMRC 1068146
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Independent Living; Disability Free Survival; Elderly; Healthy
Keywords: Survival; Functional Disability; Cardiovascular Disease; Diabetes; Dementia; Cancer
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Dementia; Neoplasms | interventions — Atorvastatin; amlodipine, atorvastatin drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Experimental): 40 mg atorvastatin (2 x 20 mg atorvastatin), taken orally once daily
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Placebo (2 x 20 mg placebo) taken orally once daily
  Interventions: Drug: Placebo (for Atorvastatin)

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 20 mg tablet
  Other Names: Lipitor, , , Cadivast, Caduet, Lorstat, Torvastat, Trovas; Atorachol; Cadatin
  Arms: Atorvastatin
Drug: Placebo (for Atorvastatin) — Inactive pill manufactured to mimic Atorvastatin 20 mg tablet
  Other Names: no other names
  Arms: Placebo

SUMMARY:
The STAREE study will examine whether treatment with statin (atorvastatin 40mg) compared with placebo will prolong disability free survival and reduce major cardiovascular events amongst healthy elderly people (≥70 years).

DETAILED DESCRIPTION:
Statin therapy has been shown to reduce the risk of vascular events in younger individuals with manifest atherosclerotic disease or at high risk of vascular events. However, data derived from meta-analyses of existing trials suggests that the efficacy of statins may decline sharply amongst those over 70-75 years of age. Insufficient patients of this age group have been included in major trials to be certain of the benefit. Within this age group part of the benefit of statin therapy may be offset by adverse effects including myopathy, development of diabetes, cancer and cognitive impairment, all of which are more prevalent in the elderly in any event.

The use of statins in the over 70 age group raises fundamental questions about the purpose of preventive drug therapy in this age group. When a preventive agent is used in the context of competing mortality, polypharmacy and a higher incidence of adverse effects its use should be justified by an improvement in quality of life or some other composite measure that demonstrates that the benefit outweighs other factors.

STAREE will determine whether taking daily statin therapy (40 mg atorvastatin) will extend the length of a disability-free life, determined from survival outside permanent residential care, in healthy participants aged 70 years and above.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥70 years living independently in the community
* Willing and able to provide informed consent and accept the study requirements (Note: competent physical ability to participate in the trial is assessed using the KATZ ADL questionnaire)

Exclusion Criteria:

A history of cardiovascular disease (defined as myocardial infarction, stroke, peripheral vascular disease, angina, transient ischaemic attack, coronary artery angioplasty and/or stenting, coronary artery bypass grafting, carotid stenosis, abdominal aortic aneurysm or heart failure),

* A history of dementia or a 3MS score <78 on screening,
* A history of diabetes,
* Total cholesterol >7.5 mmol/L,
* Moderate or severe chronic kidney disease (persistent proteinuria (Urine albumin:creatinine ratio >30mg/mmol or Urine protein:creatinine ratios >45 mg/mmol)45 and/or eGFR <45ml/min/1.73m2),
* Moderate or severe liver disease (persistent elevations of transaminases of more than 3 times the upper limit of the normal laboratory reference range),
* Serious inter-current illness likely to cause death within the next 5 years such as terminal cancer or obstructive airways disease,
* Current participation in a clinical trial,
* Absolute contraindication to statin therapy,
* Current use of statin therapy or other lipid lowering therapy for primary prevention and unwilling to stop therapy,
* Current long term or permanent use of the following cytochrome P450 (CYP) 3A4 inhibitors : Amiodarone, Boceprevir, Cimetidine, Cyclosporin, Danazol, Fosamprenavir, Indinavir, Lopinavir + Ritonavir, Erythromycin, Fluconazole, Itraconazole, Ketoconazole.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 9971 (Actual)
Dates: Start 2015-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disability free survival - death or development of dementia or development of persistent physical disability | Time from randomisation to a primary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Defined as survival free of dementia or persistent physical disability (as derived from the endpoints of all-cause mortality, dementia and physical disability)
Major cardiovascular events | Time from randomisation to a primary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Defined as the first occurrence of a cardiovascular death or a non-fatal myocardial infarction or stroke or coronary revascularisation

SECONDARY OUTCOMES:
A composite of cardiovascular death, non-fatal myocardial infarction or non-fatal stroke | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  A composite of cardiovascular death, non-fatal myocardial infarction or non-fatal stroke
Cardiovascular death | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Fatal cardiovascular events
Fatal and Non-fatal Mycocardial infarction | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Fatal and non-fatal
Hospitalisations | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Hospitalisation reasons and length of stay
Fatal and Non-fatal Cancer | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Fatal and Non-fatal Cancer (excluding non-melanoma skin cancer)
Other cognitive impairment | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Cognitive decline as assessed using cognitive tests excluding depression
Quality of life measured by the Short Form Health Survey (SF-36) | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Quality of life (measured by the Short Form Health Survey (SF-36) administered at every second year of follow-up).
Cost-effectiveness of statin | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Cost-effectiveness of statin
Fatal and Non-fatal Stroke | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Fatal and Non-fatal Stroke can be a) haemorrhagic or b) thromboembolic
Approved need for permanent residential care | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  ACAS report
Dementia | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  All-cause dementia (COWAT, Stroop test, Trail Making Test, HVLT-R, SDMT, ADAS-Cog, Lurian overlapping figures) or external diagnosis
Persistent physical disability | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  KATZ-ADL administered every 6 months or external diagnosis
All cause death | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  All cause death
Heart failure | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Heart failure
Atrial fibrillation | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Atrial fibrillation
Revascularisation procedure | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  Revascularisation procedure including coronary revascularisation

OTHER OUTCOMES:
New onset diabetes | Time from randomisation to a secondary endpoint or censoring at the end of study follow-up which is anticipated to be an average 6 years.
  New diagnosis of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Zoungas, MBBS, FRACP, Principal Investigator — Monash University
Locations (6):
- Australia (6):
  - Tasmania, Hobart, Tasmania
  - Victoria, Melbourne, Victoria
  - South Australia, Adelaide, Western Australia
  - Queensland, Brisbane
  - New South Wales, Newcastle
  - Western Australia, Perth

IPD SHARING:
Plan to Share IPD: No
On completion of the trial, and after publication of the primary and secondary outcomes of the study, requests for access to de-identified data (to be provided through a secure online environment) may be submitted to the researchers located at the School of Public Health and Preventive Medicine, Monash University, Melbourne, Australia

REFERENCES:
- [Derived] Zoungas S, Moran C, Curtis AJ, Spark S, Flanagan Z, Beilin L, Chong TT, Cloud GC, Hopper I, Kost A, McNeil JJ, Nicholls SJ, Reid CM, Ryan J, Tonkin AM, Ward S, Wierzbicki AS, Wolfe R, Zhou Z, Nelson MR; STAREE investigator group. Baseline Characteristics of Participants in STAREE: A Randomized Trial for Primary Prevention of Cardiovascular Disease Events and Prolongation of Disability-Free Survival in Older People. J Am Heart Assoc. 2024 Nov 19;13(22):e036357. doi: 10.1161/JAHA.124.036357. Epub 2024 Nov 15. PMID 39548016
- [Derived] Zoungas S, Curtis A, Spark S, Wolfe R, McNeil JJ, Beilin L, Chong TT, Cloud G, Hopper I, Kost A, Nelson M, Nicholls SJ, Reid CM, Ryan J, Tonkin A, Ward SA, Wierzbicki A; STAREE investigator group. Statins for extension of disability-free survival and primary prevention of cardiovascular events among older people: protocol for a randomised controlled trial in primary care (STAREE trial). BMJ Open. 2023 Apr 3;13(4):e069915. doi: 10.1136/bmjopen-2022-069915. PMID 37012015
- [Derived] Rozing MP, Westendorp RGJ. Altered cardiovascular risk pattern of LDL cholesterol in older adults. Curr Opin Lipidol. 2023 Feb 1;34(1):22-26. doi: 10.1097/MOL.0000000000000859. Epub 2022 Nov 16. PMID 36413436